CLINICAL TRIAL: NCT06592742
Title: The Impact of Integrating Progressive Muscle Relaxation Into Pulmonary Rehabilitation on Quality of Life, Mental Health, and Physical Function in Adults With Cystic Fibrosis: A Randomized Controlled Trial
Brief Title: Progressive Muscle Relaxation in Pulmonary Rehab for Quality of Life, Mental Health, and Sleep in Cystic Fibrosis
Acronym: PRIME-CF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spitalul Clinic de Boli Infecțioase și Pneumoftiziologie Dr. Victor Babeș Timișoara (Other Government)
Responsible Party: Principal Investigator, Crisan Alexandru Florian, Principal Investigator, Spitalul Clinic de Boli Infecțioase și Pneumoftiziologie Dr. Victor Babeș Timișoara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4989
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Cystic Fibrosis (CF)
Keywords: cystic fibrosis; mental health; sleep quality; anxiety and depression; progressive muscle relaxation
MeSH Terms: conditions — Cystic Fibrosis; Psychological Well-Being; Sleep Initiation and Maintenance Disorders; Anxiety Disorders; Depression | interventions — Single Person

STUDY DESIGN:
Intervention Model Description: In our study participants are randomly assigned to one of two groups:
  Intervention Group: receives the pulmonary rehabilitation program with PMR. Control Group: receives the standard PR program only, without PMR.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (PR alone) (Active Comparator): The control group in this study will undergo a standard pulmonary rehabilitation (PR) program designed to improve lung function, physical endurance, and overall quality of life in patients with cystic fibrosis (CF). The intervention will last for 21 days, with participants attending daily sessions of structured PR. This group will not receive the progressive muscle relaxation (PMR) component.
  Interventions: Behavioral: Pulmonary rehabilitation (alone)
- Intervention group (PR + PMR) (Experimental): The intervention group in this study will participate in the standard pulmonary rehabilitation (PR) program, similar to the control group, but with progressive muscle relaxation (PMR) sessions aimed at improving mental health, reducing anxiety, and enhancing sleep quality. This group will receive both physical and mental health interventions over the 21-day program to assess the combined impact of PR and PMR on quality of life, mental health, sleep quality, and physical endurance.
  Interventions: Behavioral: Intervention group (PR + PMR)

INTERVENTIONS:
Behavioral: Pulmonary rehabilitation (alone) — The Pulmonary Rehabilitation (PR) program for the control group includes daily aerobic exercises such as treadmill walking or cycling for 20-30 minutes at moderate intensity, tailored to improve cardiovascular fitness and respiratory function. Strength training focuses on major muscle groups with resistance exercises lasting 15-20 minutes, promoting muscle strength and endurance. Airway clearance techniques are performed for 15-20 minutes daily, using methods like chest physiotherapy or positive expiratory pressure (PEP) to clear mucus from the lungs. Breathing exercises, including diaphragmatic and pursed-lip breathing, are practiced for 10-15 minutes to improve breathing efficiency. Participants also receive education on disease management and nutritional support to meet caloric needs.
  Other Names: PR
  Arms: Control group (PR alone)
Behavioral: Intervention group (PR + PMR) — The intervention group will follow a Pulmonary Rehabilitation (PR) program combined with Progressive Muscle Relaxation (PMR). Daily aerobic exercises like treadmill walking or cycling will be performed for 20-30 minutes at moderate intensity, improving cardiovascular fitness and lung function. Strength training for major muscle groups will be included, with 15-20 minutes of resistance exercises to enhance muscle strength. Airway clearance techniques, such as chest physiotherapy or PEP, will help clear mucus from the lungs in daily 15-20 minute sessions. Breathing exercises, including diaphragmatic and pursed-lip breathing, will be practiced for 10-15 minutes to improve breathing efficiency. The PMR component involves daily 20-30 minute guided sessions to reduce stress and anxiety through muscle relaxation techniques.
  Other Names: PMR
  Arms: Intervention group (PR + PMR)

SUMMARY:
This study, called PRIME-CF, will look at how adding progressive muscle relaxation (PMR) to a typical pulmonary rehabilitation (PR) program might help adults with cystic fibrosis (CF). CF is a long-term disease that affects the lungs and can cause physical and mental health challenges, including anxiety, depression, and trouble sleeping.

The study will involve two groups: one group will follow the usual PR program, which includes exercises to improve lung function and overall health, while the other group will also practice PMR, a technique to help relax muscles and reduce stress. The main goal is to see if adding PMR can improve participants quality of life, reduce anxiety and depression, and improve sleep quality.

Investigators will use questionnaires to measure how participants feel about their mental and physical health and tests to assess their physical endurance, such as measuring how far they can walk in six minutes (6-Minute Walk Test).

Investigators hope to find a better way to support people with CF in managing their physical and emotional health by combining physical therapy with relaxation techniques.

DETAILED DESCRIPTION:
Our study aims to evaluate the effects of integrating progressive muscle relaxation (PMR) into a standard pulmonary rehabilitation (PR) program on quality of life, mental health, sleep quality, and physical endurance in adults with cystic fibrosis (CF). CF is a chronic genetic disorder that imposes a heavy physical and psychological burden on patients, often resulting in anxiety, depression, and sleep disturbances. While PR effectively improves lung function and physical capacity, its impact on mental health and sleep quality is less established. PMR, a relaxation technique that reduces stress and improves mental well-being, is integrated into this study's PR program to assess whether it can further enhance outcomes in CF patients.

The study will include adults with CF randomly assigned to either a control group (standard PR program) or an intervention group (PR program plus PMR). The PR program will involve daily exercise sessions, including aerobic and strength training, airway clearance techniques, and medical education. The intervention group will also participate in daily guided PMR sessions designed to reduce muscle tension and psychological stress.

The studys primary outcomes will be changes in quality of life, assessed using the Cystic Fibrosis Questionnaire-Revised (CFQ-R), and mental health, measured by the Hospital Anxiety and Depression Scale (HADS). Secondary outcomes include improvements in sleep quality, measured by the Pittsburgh Sleep Quality Index (PSQI), and physical endurance, assessed via the 6-Minute Walk Test (6MWT). Data will be collected at baseline, post-intervention, and at a 4-week follow-up to evaluate the sustainability of any benefits.

The study is designed to determine whether adding PMR to a PR program can meaningfully improve CF management in both the physical and mental health domains, offering a more comprehensive approach to the care of adult CF patients. The findings are expected to contribute to developing more holistic treatment protocols for CF, integrating mental health interventions into traditional pulmonary rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed cystic fibrosis diagnosis based on clinical, genetic, or sweat chloride testing, as defined by established CF diagnostic criteria.
* 18 years or older at the time of enrollment
* Participants must have stable lung function, defined as a Forced Expiratory Volume in 1 second (FEV1)
* Participants must not have had a pulmonary exacerbation requiring hospitalization or intravenous (IV) antibiotics within the past 4 weeks before the start of the study
* Physically able to engage in the daily exercise and airway clearance components of the pulmonary rehabilitation program
* Participants must be willing and able to participate in daily progressive muscle relaxation
* Participants must be on a stable medication regimen for at least 4 weeks before study enrollment
* Participants must be non-smokers or have quit smoking for at least 6 months before enrollment
* Participants must be able to understand and provide written informed consent, indicating their willingness to participate in the study, adhere to the intervention schedule, and comply with follow-up assessments

Exclusion Criteria:

* Participants who have experienced a pulmonary exacerbation or acute respiratory infection requiring hospitalization or intravenous (IV) antibiotics within the last 4 weeks
* Participants who have undergone a lung transplant or any other major surgery within the past 6 months
* Participants with severe comorbid conditions such as: uncontrolled cardiovascular disease, renal or liver failure, severe musculoskeletal disorders, severe or uncontrolled psychiatric disorders
* Participants who have had significant changes in their medication regimen within the last 4 weeks
* Participants with uncontrolled diabetes

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2024-09-13 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Health related Quality of life | At inclusion, at 21 days, at 48 days.
  The Cystic Fibrosis Questionnaire-Revised (CFQ-R) is a disease-specific tool designed to assess the health-related quality of life in individuals with cystic fibrosis (CF). It includes 47 items that cover several domains: physical functioning, emotional well-being, vitality, social functioning, body image, eating problems, treatment burden, respiratory symptoms, and digestive symptoms. Scores range from 0 to 100, with higher scores indicating better quality of life. The CFQ-R is used in clinical trials, research, and routine care to measure the impact of CF on daily life and the effectiveness of interventions.
Mental Health | At inclusion, at 21 days, at 48 days.
  The Hospital Anxiety and Depression Scale (HADS) is a widely used tool to assess symptoms of anxiety and depression in patients with physical health conditions. It consists of 14 items, divided into two subscales: 7 for anxiety (HADS-A) and 7 for depression (HADS-D). Each item is scored on a scale from 0 to 3, with total scores ranging from 0 to 21 for each subscale. Higher scores indicate greater levels of anxiety or depression. Scores are categorized as normal (0-7), mild (8-10), moderate (11-14), or severe (15-21).

SECONDARY OUTCOMES:
Sleep Quality | At inclusion, at 21 days, at 48 days.
  The Pittsburgh Sleep Quality Index (PSQI) is a widely used tool designed to assess sleep quality and identify sleep disturbances over a 1-month period. It consists of 19 self-rated items that are grouped into seven components: sleep duration, sleep latency, sleep efficiency, sleep disturbances, use of sleep medication, daytime dysfunction, and subjective sleep quality. Each component is scored from 0 to 3, with a total score ranging from 0 to 21; higher scores indicate worse sleep quality. A total score above 5 suggests poor sleep quality.
Physical Endurance | At inclusion, at 21 days, at 48 days.
  The 6-Minute Walk Test (6MWT) is a simple, practical test used to assess functional exercise capacity in patients with chronic conditions, including cystic fibrosis. During the test, a patient walks for 6 minutes on a flat, straight course, aiming to cover as much distance as possible at their own pace, while taking breaks if necessary. The total distance walked, measured in meters, is the main outcome, with a longer distance indicating better exercise capacity.
Lung Function | At inclusion, at 21 days, at 48 days.
  Lung function will assess the impact of the intervention (PR + PMR) on participants respiratory health. The primary tool used for this evaluation will be spirometry. This standard pulmonary function test measures how well the lungs work by assessing the volume and flow of air during breathing. Forced Expiratory Volume in 1 Second (FEV1) will be recorded. It reflects airway obstruction, with improvements indicating better lung function. FEV1 is reported as a percentage of the predicted value based on age, sex, and height.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandru Crisan, Phd, Principal Investigator — University of Medicine and Pharmacy "Victor Babes" Timisoara
Locations (1):
- Hospital of Infectious Disease and Pneumoftiziology Victor Babes, Timișoara, Romania

IPD SHARING:
Plan to Share IPD: No